CLINICAL TRIAL: NCT04334200
Title: The Development and Evaluation of a Culturally Tailored Support Group Program on the Psychosocial Wellbeing of Family Caregivers of Individuals Living With Dementia in Hong Kong
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Yiu Hing Cheung, PhD student (Nursing), Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019.565
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Intervention group receiving support group program
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cultivate yourself: support for caregivers of dementia persons (Experimental): There will be six sessions (1 or 2 session per week). The duration of each session will be 1.5-2 hours per session. The contents include: introduction on dementia, caregivers' role, how to communicate with dementia persons, tips on caregiving, stress and emotional management. The training content has been verified by one social worker, family caregivers of individuals living with dementia and a teacher who teach Chinese, Chinese history and culture in the secondary school in Hong Kong. No adverse comments are received from them.
  Interventions: Behavioral: Cultivate yourself: support for caregivers of dementia persons

INTERVENTIONS:
Behavioral: Cultivate yourself: support for caregivers of dementia persons — The Chinese cultural values, including philosophical thoughts, will be included in the intervention. Chinese philosophical thoughts including the concepts of moderation, improving oneself, and harmony with nature will be used in the intervention. Confucianism, Taoism and Buddhism are the foundation for Chinese for concepts of health and illness, health promotion, and health-seeking behavior. Therefore, it is necessary to incorporate such philosophies in the sessions of the program.

SUMMARY:
Hong Kong is also facing the increasing prevalence of dementia. Evidence states that dementia caregivers have poor psychosocial wellbeing including stress, depression and anxiety. Effective services and interventions should be provided to the caregivers to improve their psychosocial wellbeing. Recent studies suggest that cultural adapted intervention is necessary. Such intervention can support caregivers to improve psychosocial wellbeing by using the culture and rituals to relevant racial caregivers creatively. Among all interventions for dementia caregivers, it was reported that the support group/program was more effective to improve psychosocial well-being of dementia caregivers. However, the studies about support group for dementia caregivers did not report the cultural sensitivity elements explicitly. Most of them mention the component 'language' only. Other elements, including philosophical thoughts, had not been mentioned in the articles. It is necessary to provide more cultural components including philosophical thoughts in the support groups. Moreover, the studies did not report on the benefits of adding cultural elements in the interventions to dementia caregivers. Although the literature mentioned cultural adapted interventions were beneficial, the research on understanding its benefits is inadequate. More caregiver intervention studies to understand the advantages of cultural tailoring are needed. Hence, we need to do more studies to understand the benefits of adding cultural elements in the interventions to caregivers. A research is performed to develop and evaluate a culturally adapted intervention for dementia caregivers to improve their psychosocial wellbeing.

This research study is to evaluate the effectiveness and benefits of culturally tailored interventions for caregivers of older adults with dementia on improving psychosocial well-being. Mixed method and quasi-experimental design will be applied. There are 2 groups: intervention and control groups. Each group needs to complete pre and post-test to assess their psychosocial well-beings. The pre and post-test data will be used for assessing the effectiveness of the culturally tailored intervention program for the dementia caregivers. For intervention group, qualitative data, i.e. data from focus group interview will be performed to assess the benefits of inclusion of cultural elements in the program.

DETAILED DESCRIPTION:
A quasi-experimental study will be performed to assess the effectiveness and benefits of a culturally tailored support group programs for Chinese dementia caregivers. The PhD candidate will contact three non-governmental organizations (NGO), including Rotary Club that provides dementia services to dementia persons or their caregivers in the elderly centres. The caregivers will be recruited as participants through these centres.

A quasi-experimental, non-equivalent pre-test-post-test control group design will be used to determine the effectiveness of a culturally tailored support group program. A non-equivalent control group design was used because caregivers from the same centre would have known each other. If caregivers in each elderly centre were randomly assigned to experimental and control groups, there may have been a chance that caregivers in the experimental group would discuss the intervention with caregivers in the control group. Also, the caregivers in the control group may think it was unfair that they do not have a chance to have the culturally tailored support group programs. Hence, a quasi-experimental design will be implemented and the experimental and control groups will be from different elderly centres.

The participants should be the family members who care for a relative with dementia at home. The eligibility criteria include:

1. Chinese;
2. aged > 18 years;
3. the ability to communicate in Chinese / Cantonese; and
4. voluntary participation. The exclusion criteria include those currently suffering from a psychiatric illness with/without regular follow-up or treatment.

ELIGIBILITY:
Inclusion Criteria:

* The participants should be the family members who care for a relative with dementia at home. The eligibility criteria include:

  1. Chinese;
  2. aged > 18 years;
  3. the ability to communicate in Chinese / Cantonese; and
  4. voluntary participation.

Exclusion Criteria:

* The exclusion criteria include those currently suffering from a psychiatric illness with/without regular follow-up or treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
SSQ6 | 1.5 month
  • The SSQ6 was used to investigate the quantity of support each participant obtains as well as their satisfaction with the support provided. The participants will be asked to indicate from 0-9 the number of support persons they have for the six situations and rate their overall satisfaction with the support provided using a six-point scale. High SSQ6 satisfaction scores mean more satisfaction with social support received.